CLINICAL TRIAL: NCT03066219
Title: A Multi-Center, Randomized, Double Masked, Placebo Controlled Clinical Study to Assess the Safety and Efficacy of BRM421 Ophthalmic Solution in Subjects With Dry Eye Using a Controlled Adverse Environment (CAE®) Model
Brief Title: Safety and Efficacy of BRM421 for Dry Eye Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BRIM Biotechnology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRM421-16-C001-PR
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BRM421 Ophthalmic Solution (Active Comparator): The active control with BRM421 solution
  Interventions: Drug: BRM421
- Placebo (Placebo Comparator): The vehicle solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BRM421 — A topical solution of BRIM421 ophthalmic drops
  Arms: BRM421 Ophthalmic Solution
Drug: Placebo — vehicle ophthalmic drops
  Arms: Placebo

SUMMARY:
The objective of this study is to compare the safety and efficacy of BRM421 Ophthalmic Solution to placebo for the treatment of the signs and symptoms of dry eye.

DETAILED DESCRIPTION:
This is a multi-center, double-masked, randomized, vehicle-controlled, phase 2 study in approximately 150 subjects. (75 per treatment arm).

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent;
* Have a reported history of dry eye for at least 6 months prior to enrollment;
* Have a history of use of eye drops

Exclusion Criteria:

* Have any clinically significant slit lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction (MGD), lid margin inflammation or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters;
* Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1;
* Have worn contact lenses within 7 days of Visit 1 or anticipate using contact lenses during the study;
* Have used any eye drops within 2 hours of Visit 1;
* Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months;
* Be a woman of childbearing potential who is not using an acceptable means of birth control; acceptable methods of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2017-05-20 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Sign: Corneal fluorescein staining score | Up to 4 weeks
Symptom: Ocular discomfort score | Up to 4 weeks

SECONDARY OUTCOMES:
Tear film break-up time | Up to 4 weeks
Conjunctival Redness | Up to 4 weeks
Ocular Surface Disease Index (OSDI)© | Up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Central Maine Eye Care, Lewiston, Maine
  - Andover Eye Associates, Andover, Massachusetts